CLINICAL TRIAL: NCT03921567
Title: Intravenous Lidocaine for Perioperative and Postoperative Analgesia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rajmonda Nallbani-Komoni (Other)
Responsible Party: Sponsor-Investigator, Rajmonda Nallbani-Komoni, Principal investigator, University Clinical Centre of Kosova
Organization: University Clinical Centre of Kosova (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: UCCKosovo
Record Dates: First submitted 2019-04-16; First posted 2019-04-19 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Analgesic Drug Dependence
Keywords: Analgesia; Perioperative periode; Postoperative periode; VAS scale
MeSH Terms: conditions — Agnosia | interventions — Lidocaine; Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group I (Experimental): at induction of anesthesia will be given lidocaine 2mg / kg / i.v., bolus, and in perioperative and postoperative period will be given lidocaine 1.5mg / kg / h-1, continuously during surgery and 48 hours after surgery.
  Interventions: Drug: Lidocaine Hydrochloride
- Group II (Active Comparator): at induction of anesthesia will be given lidocaine 2mg / kg / i.v., bolus, and ketamine 0.15mg / kg / , bolus, i.v .; lidocaine will continue during the operation and in the postoperative period with a dose of 1.5mg / kg / h-1, continuously, during the operation and 48 hours after the operation
  Interventions: Drug: Lidocaine Hydrochloride; Drug: Lidocaine Hydrochloride and Ketamine
- The control group (Placebo Comparator): will be given opioids during surgery, opioids and nonsteroid antiinflammatory agents will be given 48 hours after surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine Hydrochloride — at induction of anesthesia will be given lidocaine 2mg / kg / i.v., bolus, and in perioperative and postoperative period will be given lidocaine 1.5mg / kg / h-1, continuously during surgery and 48 hours after surgery.
  Other Names: Lidocaine Hydrochloride ampule
  Arms: Group I; Group II
Drug: Lidocaine Hydrochloride and Ketamine — at induction of anesthesia will be given lidocaine 2mg / kg / i.v., bolus, and ketamine 0.15mg / kg / , bolus, i.v .; lidocaine will continue during the operation and in the postoperative period with a dose of 1.5mg / kg / h-1, continuously, during the operation and 48 hours after the operation
  Other Names: Lidocaine Hydrochloride ampule and Ketamine ampule
  Arms: Group II
Drug: Placebo — will be given opioids during surgery, and opioids and nonsteroid antiinflammatory agents will be given 48 hours after surgery.
  Other Names: Placebo for(lidocaine hydrochloride)
  Arms: The control group

SUMMARY:
Postoperative pain continues to be untreated despite the application of multimodal analgesia, medication and new analgesic techniques. Traditional opioid pain treatment has many side effects, while invasive methods, such as epidural catheter, have high costs and difficulties during application.

Lidocaine is a local anesthetic and its administration with intravenous routes has analgesic, antihyperalgic and antiinflammatory action. It increases the motility of the intestine and has antiemetic properties. The advantage of this method is the low cost of the preparation and its easy application. The intravenous administration of lidocaine for postoperative analgesia is recently used and not sufficiently researched technique .

DETAILED DESCRIPTION:
The purpose of this research is to investigate the analgesic effects of intravenous lidocaine in the perioperative and postoperative period, on various surgical interventions. In the perioperative period, its effect on the reduction of opiodic use will be evaluated, while during the postoperative period will be evaluate the degree of analgesia, the rate of reduction of additional analgesics, the impact on the clinical parameters and the patient's rehabilitation.

The research will be conducted at the Clinic of Gynecology and Obstetrics, the Surgery Clinic, the Urology Clinic, the Orthopedic Clinic, of Universitary Clinical Centre of Kosovo and the American Hospital in Pristina, Republic of Kosovo.

The study will be conducted during the period April 2018 - January 2020.

After obtaining a permit from the ethics committee, all patients to be investigated will be informed first through the information form for all the risks and advantages of this analgesic technique and from them will be consented to their participation in the research.

In the intervention group of the study will be included 520 patients of both genders and ages 18-65 years. Patients will undergo these surgical interventions: gynecological, abdominal, laparoscopical, urological and orthopedic interventions.

The intervention group includes two groups for each type of surgery:

Group I (n = 50); at induction of anesthesia will be given lidocaine 2mg / kg / i.v., bolus, and in perioperative and postoperative period will be given lidocaine 1.5mg / kg / h-1, continuously during surgery and 48 hours after surgery.

Group II (n = 50); at induction of anesthesia will be given lidocaine 2mg / kg / i.v., bolus, and ketamine 0.15mg / kg / , bolus, i.v .; lidocaine will continue during the operation and in the postoperative period with a dose of 1.5mg / kg / h-1, continuously, during the operation and 48 hours after the operation.

The control group (n = 30) will be given opioids during surgery, and opioids and nonsteroid antiinflammatory agents will be given 48 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age of both genders from 18 to 75 years
* ASA physiological status I-III
* Participation in abdominal, orthopedic, laparoscopical, gynecological and urological interventions.

Exclusion Criteria:

* Patient rejection
* History of chronic opioid intake
* History of renal, hepatic or psychiatric disorders
* Heart failure,
* Organ transplant history,
* Lidocaine allergy
* Family history of malignant hyperthermia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-10-30 (Estimated); Study Completion 2020-01-30 (Estimated)

PRIMARY OUTCOMES:
Reduction of opiods used during perioperative period and other analgesics used during postoperative period | 48 hours after surgical intervention
  The primary outcome measures are: the use of opiods and other analgesics during and 48 hours after the surgical intervention.
  During the intraoperative period, it will be investigated how the application of intravenous lidocaine will reduce the amount of opiodes used, amd during the postoperative period will be investigated when the application of other analgesics will start and which analgesics will be used as well,how often they will be given and in which dose.
  The analgesics which will be investigated include routine analgesics found in our hospital:
  * tramadol
  * acetaminophen
  * diclophenac
  * ketorolac
  * others

SECONDARY OUTCOMES:
Pain scores measured at rest and during the movement with Visual Analog Scale | 48 hours after surgical intervention
  * Pain scores measured at rest and during the movement with Visual Analog Scale
  * the beginning of the intestinal motility,
  * side effects (nausea, vomiting, headache, hypotension, arrhythmias, dizziness ,hallucinations etc)
  Postoperative analgesia will be determined through the VAS scale-Visual Analog Scale. This scale will be used to determinate the intensity of pain in patients in the postoperative period, initially determining the intensity of pain in silence as well as after mobilization or motion, i.e Visual Dynamic Scale.
  This scale determines the intensity of the pain and is expressed in a numeric value from1-10. 0- no pain, 1-2- mild pain, 3-6 moderate pain, 7-10 severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Antigona Hasani, Profesor, Study Director — University of Pristina, Faculty of Medicine, 10000 Pristina, Kosovo
Locations (2):
- Kosovo (2):
  - University Clinical Centre of Kosovo, Pristina
  - University of Pristina, Faculty of Medicine, Pristina

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data for primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion
Access Criteria: Requestors will be required to sign a Data Access Agreement and then these requests will be reviewed by an Independent Review Panel.

REFERENCES:
- [Background] 1. Mendonça* FT, Reis MC, Aguiar JA and Calvano LA Systemic Lidocaine for Perioperative Analgesia: A Literature Review, J Anest & Inten Care Med. 2015;1(1): 555551.
- [Result] Apfelbaum JL, Chen C, Mehta SS, Gan TJ. Postoperative pain experience: results from a national survey suggest postoperative pain continues to be undermanaged. Anesth Analg. 2003 Aug;97(2):534-540. doi: 10.1213/01.ANE.0000068822.10113.9E. PMID 12873949
- [Result] Tanaka PP, Moss J. The role of peripheral opiate antagonists in pain medicine and perioperative care. Rev Bras Anestesiol. 2008 Sep-Oct;58(5):540-7, 533-9. doi: 10.1590/s0034-70942008000500011. English, Portuguese. PMID 19382412
- [Result] de Oliveira CM, Issy AM, Sakata RK. Intraoperative intravenous lidocaine. Rev Bras Anestesiol. 2010 May-Jun;60(3):325-33. doi: 10.1016/S0034-7094(10)70041-6. PMID 20682165
- [Result] Lauretti GR. Mechanisms of analgesia of intravenous lidocaine. Rev Bras Anestesiol. 2008 May-Jun;58(3):280-6. doi: 10.1590/s0034-70942008000300011. English, Portuguese. PMID 19378524
- [Result] McLure HA, Rubin AP. Review of local anaesthetic agents. Minerva Anestesiol. 2005 Mar;71(3):59-74. PMID 15714182
- [Result] Becker DE, Reed KL. Essentials of local anesthetic pharmacology. Anesth Prog. 2006 Fall;53(3):98-108; quiz 109-10. doi: 10.2344/0003-3006(2006)53[98:EOLAP]2.0.CO;2. PMID 17175824
- [Result] Sun Y, Li T, Wang N, Yun Y, Gan TJ. Perioperative systemic lidocaine for postoperative analgesia and recovery after abdominal surgery: a meta-analysis of randomized controlled trials. Dis Colon Rectum. 2012 Nov;55(11):1183-94. doi: 10.1097/DCR.0b013e318259bcd8. PMID 23044681
- [Result] Mao J, Chen LL. Systemic lidocaine for neuropathic pain relief. Pain. 2000 Jul;87(1):7-17. doi: 10.1016/S0304-3959(00)00229-3. PMID 10863041
- [Result] Swenson BR, Gottschalk A, Wells LT, Rowlingson JC, Thompson PW, Barclay M, Sawyer RG, Friel CM, Foley E, Durieux ME. Intravenous lidocaine is as effective as epidural bupivacaine in reducing ileus duration, hospital stay, and pain after open colon resection: a randomized clinical trial. Reg Anesth Pain Med. 2010 Jul-Aug;35(4):370-6. doi: 10.1097/AAP.0b013e3181e8d5da. PMID 20588151
- [Result] Marret E, Rolin M, Beaussier M, Bonnet F. Meta-analysis of intravenous lidocaine and postoperative recovery after abdominal surgery. Br J Surg. 2008 Nov;95(11):1331-8. doi: 10.1002/bjs.6375. PMID 18844267
- [Result] Vigneault L, Turgeon AF, Cote D, Lauzier F, Zarychanski R, Moore L, McIntyre LA, Nicole PC, Fergusson DA. Perioperative intravenous lidocaine infusion for postoperative pain control: a meta-analysis of randomized controlled trials. Can J Anaesth. 2011 Jan;58(1):22-37. doi: 10.1007/s12630-010-9407-0. PMID 21061107
- [Result] McCarthy GC, Megalla SA, Habib AS. Impact of intravenous lidocaine infusion on postoperative analgesia and recovery from surgery: a systematic review of randomized controlled trials. Drugs. 2010 Jun 18;70(9):1149-63. doi: 10.2165/10898560-000000000-00000. PMID 20518581
- [Result] Kranke P, Jokinen J, Pace NL, Schnabel A, Hollmann MW, Hahnenkamp K, Eberhart LH, Poepping DM, Weibel S. Continuous intravenous perioperative lidocaine infusion for postoperative pain and recovery. Cochrane Database Syst Rev. 2015 Jul 16;(7):CD009642. doi: 10.1002/14651858.CD009642.pub2. PMID 26184397
- [Result] Kuo CP, Jao SW, Chen KM, Wong CS, Yeh CC, Sheen MJ, Wu CT. Comparison of the effects of thoracic epidural analgesia and i.v. infusion with lidocaine on cytokine response, postoperative pain and bowel function in patients undergoing colonic surgery. Br J Anaesth. 2006 Nov;97(5):640-6. doi: 10.1093/bja/ael217. Epub 2006 Sep 4. PMID 16952918
- [Result] Kaba A, Laurent SR, Detroz BJ, Sessler DI, Durieux ME, Lamy ML, Joris JL. Intravenous lidocaine infusion facilitates acute rehabilitation after laparoscopic colectomy. Anesthesiology. 2007 Jan;106(1):11-8; discussion 5-6. doi: 10.1097/00000542-200701000-00007. PMID 17197840
- [Result] Wu CT, Borel CO, Lee MS, Yu JC, Liou HS, Yi HD, Yang CP. The interaction effect of perioperative cotreatment with dextromethorphan and intravenous lidocaine on pain relief and recovery of bowel function after laparoscopic cholecystectomy. Anesth Analg. 2005 Feb;100(2):448-453. doi: 10.1213/01.ANE.0000142551.92340.CC. PMID 15673874
- [Result] Koppert W, Weigand M, Neumann F, Sittl R, Schuettler J, Schmelz M, Hering W. Perioperative intravenous lidocaine has preventive effects on postoperative pain and morphine consumption after major abdominal surgery. Anesth Analg. 2004 Apr;98(4):1050-1055. doi: 10.1213/01.ANE.0000104582.71710.EE. PMID 15041597
- [Result] Herroeder S, Pecher S, Schonherr ME, Kaulitz G, Hahnenkamp K, Friess H, Bottiger BW, Bauer H, Dijkgraaf MG, Durieux ME, Hollmann MW. Systemic lidocaine shortens length of hospital stay after colorectal surgery: a double-blinded, randomized, placebo-controlled trial. Ann Surg. 2007 Aug;246(2):192-200. doi: 10.1097/SLA.0b013e31805dac11. PMID 17667496
- [Result] Saadawy IM, Kaki AM, Abd El Latif AA, Abd-Elmaksoud AM, Tolba OM. Lidocaine vs. magnesium: effect on analgesia after a laparoscopic cholecystectomy. Acta Anaesthesiol Scand. 2010 May;54(5):549-56. doi: 10.1111/j.1399-6576.2009.02165.x. Epub 2009 Nov 16. PMID 19919581